CLINICAL TRIAL: NCT05763407
Title: Early Feasibility Study of the NORM™ System in Heart Failure Patients (FUTURE-HFII)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Foundry Innovation & Research 1, Limited (FIRE1) (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: TF03-CID02
Record Dates: First submitted 2023-02-28; First posted 2023-03-10 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-10

CONDITIONS: Heart Failure
Keywords: Cardiovascular Disease
MeSH Terms: conditions — Heart Failure; Cardiovascular Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- NORM™ System (Experimental): NORM™ System
  Interventions: Device: NORM™ System

INTERVENTIONS:
Device: NORM™ System — NORM™ System

SUMMARY:
Early Feasibility Study of the NORM™ System in Heart Failure Patients

DETAILED DESCRIPTION:
Eligible patients who have HF and were hospitalised/treated for an episode of worsening HF within the last 12 months and/or elevated NTproBNP levels.

This non-randomised trial will enroll up to 30 patients, and the primary safety and technical endpoints will be assessed at 3 months. Safety measures will include an assessment of all adverse events. Subjects will remain in this study for 24 months.

ELIGIBILITY:
Main Inclusion Criteria

* Adults 18 years of age or older.
* Patients meeting diagnostic criteria for heart failure diagnosis for greater than 90 days and are on optimally tolerated medical therapy for at least 30 days, as recommended according to current AHA/ACC/HFSA guidelines with any intolerance or contraindications documented, regardless of ejection fraction, as evidenced by meeting either 2a, 2b, OR 2c criterion below:

  1. NYHA functional class III: with documented HF decompensation within the previous 12 months resulting in a primary HF hospitalization, HF treatment in a hospital day-care setting or unscheduled visit to a healthcare provider for administration of an intravenous diuretic to treat HF and NT-proBNP ≥600 pg/mL (or BNP ≥200 pg/mL). For patients presenting with atrial fibrillation NT-proBNP ≥900 pg/mL (or BNP ≥300 pg/mL).

     OR
  2. NYHA functional class III: NT-proBNP ≥1000 pg/mL (or BNP ≥300pg/mL). For patients presenting with atrial fibrillation NT-proBNP≥1,600 pg/mL (or BNP ≥500 pg/mL).

     OR
  3. NYHA functional class II: with documented HF decompensation within the previous 12 months resulting in a primary HFhospitalization, HF treatment in a hospital day-care setting or unscheduled visit to a healthcare provider for administration of an intravenous diuretic to treat HF AND NT-proBNP ≥1000 pg/mL (or BNP ≥300 pg/mL). For those patients presenting with atrial fibrillation NT-proBNP ≥1,600 pg/mL (or BNP ≥500 pg/mL).
* Patients must also be on a daily dose of loop diuretic of 40mg or more furosemide, or equivalent, for the 2 weeks prior to screening.
* IVC diameter within the landing zone of between 14mm and 28mm.
* Minimum IVC landing zone length of 60mm.
* Patient has sufficient Cellular and/ or Wi-Fi Internet coverage at home.
* Provide informed consent for participation in the clinical investigation and be willing and able to comply with the required daily system readings, care plan instructions, and clinical follow-up visits according to the specified schedule.

Main Exclusion Criteria:

* Significant comorbidity that, in the investigator's opinion, would results in the patient being unable to safely undergo the procedure or participate in the clinical investigation.
* Patients with an estimated Glomerular Filtration Rate (eGFR) < 25 ml/min/1.73m2
* Patients with an in vivo IVC filter, abnormal IVC or femoral venous anatomy or known congenital malformation or absence of IVC or occlusive or free-floating thrombus in the IVC.
* Patients who have severe right sided valvular disease or a right sided mechanical valve.
* Patients with a cardiac resynchronization therapy device implanted ≤ 3 months to prior to screening.
* Patients who have undergone invasive cardiac surgery in the 3 months prior to screening.
* Patients who have undergone percutaneous valve / structural heart intervention in in the 3 months prior to screening.
* Patients who have received heart transplant or a ventricular assist device or planned for advanced therapies within the next year.
* Patients with conditions associated with occlusion of the IVC, iliac or common femoral veins.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2023-06-19 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Primary Safety Endpoint - Procedural success | 30 days
  Procedural success defined as Sensor deployment at the intended site without procedural related SAEs
Primary Safety Endpoint - Freedom from Sensor Complications | 3 months
  Freedom from Sensor complications including device migration, clinically significant fracture and/or clinically significant perforation of the Inferior Vena Cava (IVC) or symptomatic caval thrombosis
Primary Effectiveness Endpoint - Device Performance | 3 months
  Device performance defined as an assessment of the ability of the NORM™ System to successfully transmit collected data to a secure database

SECONDARY OUTCOMES:
Exploratory Safety Outcome | 24 months
  Summary of all device / system related adverse events (AEs)
Exploratory Safety Outcome | 24 months
  Summary of all device / system related complications

CONTACTS AND LOCATIONS:
Overall Officials: Carolyn Borme, Study Director — Director Clinical US
Locations (8):
- United States (8):
  - University of Minnesota Medica Center, Minneapolis, Minnesota
  - Columbia University Irving Medical Center/ New York Presbyterian Hospital, New York, New York
  - Rochester General Hospital, Rochester, New York
  - Duke University Medical Center, Durham, North Carolina
  - Cleveland Clinic, Cleveland, Ohio
  - The Ohio State University Wexner Medical Center, Columbus, Ohio
  - Prisma Health, Greenville, South Carolina
  - Austin Heart Central at the Heart Hospital of Austin, Austin, Texas

IPD SHARING:
Plan to Share IPD: No